CLINICAL TRIAL: NCT06533709
Title: Satisfactory Debulking Prediction Model for Advanced Ovarian Cancer Based on PET-CT Image Data and Its Clinical Application
Brief Title: Satisfactory Debulking Prediction Model for Advanced Ovarian Cancer Based on PET-CT Image Data
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-503-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer; Image; Predation
Keywords: Ovarian Cancer; PET-CT Image; Debulking Prediction Model
MeSH Terms: conditions — Ovarian Neoplasms; Predatory Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SYSU cohort: Patients cohort from Sun Yat-sen Memorial Hospital, as the training cohort.
  Interventions: Diagnostic Test: Radio-score
- ZJCH cohort: Patients cohort from Zhejiang Cancer Hospital, as the external validation cohort.
  Interventions: Diagnostic Test: Radio-score

INTERVENTIONS:
Diagnostic Test: Radio-score — A score based on the LASSO regression model predicting the R0 resection of the primary debulking surgery of advanced ovarian cancer.

SUMMARY:
This project intends to conduct a multicenter retrospective study to evaluate the satisfactory reduction of advanced ovarian cancer using PET-CT images, and explore the correlation between molecular biological characteristics and clinical characteristics of ovarian cancer through high-throughput sequencing genomics combined with radiomics.

DETAILED DESCRIPTION:
Ovarian cancer is the gynecological malignant tumor with the highest fatality rate. More than 70% of patients are diagnosed with advanced stage, often involving various organs of the pelvis and abdomen, which increases the difficulty of surgical resection, and the 5-year survival rate is only 30%. Surgical treatment is the cornerstone of the treatment of ovarian cancer, and whether it can achieve satisfactory tumor reduction is an important factor affecting the prognosis of ovarian cancer. At present, the methods used to evaluate whether satisfactory tumor reduction can be achieved include Suidan score based on CT image and Fagotti score based on laparoscopic exploration, but there are problems such as low sensitivity, poor specificity or strong subjectivity, and the efficiency of predicting satisfactory tumor reduction is only about 60%. In recent years, PET-CT has been widely used in tumor diagnosis. Pet-ct combined with PET metabolic imaging technology and traditional CT scanning can help to distinguish the nature of tumors, assess the systemic tumor load, define the scope of the lesion, and provide the metabolic status of various parts of the body. The application value of PET-CT related imaging features and metabolic information in ovarian cancer needs to be clarified. Our team's previous study found that PET-CT related images and metabolic information showed certain advantages in predicting satisfactory resection of ovarian cancer, and the AUC reached 0.85, which was better than the current CT image score and laparoscopic score. Therefore, this project intends to conduct a multicenter retrospective study to evaluate the satisfactory tumor reduction rate of advanced ovarian cancer using PET-CT images to guide clinical practice and predict the prognosis of patients. At the same time, we will explore the molecular biological characteristics and clinical relevance of ovarian cancer through the combination of high-throughput sequencing genomics and radiomics.

ELIGIBILITY:
Inclusion Criteria:

* Pathological type is epithelial ovarian cancer.
* Underwent primary debulking surgery at our hospital.
* Postoperative pathological staging is FIGO stage IIB or above.
* Clinical, surgical, and pathological data of the patient are mostly complete.

Exclusion Criteria:

* Pathological type is non-epithelial ovarian cancer.
* Underwent fertility-preserving surgery or palliative surgery.
* Presence of infection during PET/CT image acquisition.
* Concurrent other malignant tumors.
* Severe diseases of other major organs.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 96 patients with advanced ovarian cancer who underwent PET-CT examination before the surgery, and received primary debulking surgery at our center from July 2017 to April 2024 were included for model development. Additionally, 50 patients from Zhejiang Cancer Hospital were included for model validation.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection | yes or not
  In patients with advanced ovarian cancer, the residual status after initial cytoreductive surgery is defined as follows: complete resection is defined as R0 resection, whereas visible residual tumor lesions during surgery are defined as non-R0 resection

SECONDARY OUTCOMES:
5-year progression-free survival (PFS) | 5 years
  PFS was calculated from the date of the last chemotherapy until disease progression or death due to any cause.
5-year overall survival (OS) | 5-year
  OS was calculated from the date of the primary debulking surgery until death due to any cause.
Response to platinum-based chemotherapy | At least 6 months after the last chemotherapy
  After the last chemotherapy, treatment efficacy was assessed according to NCCN guidelines. For primary tumor, patients who relapsed 6 months or more after initial chemotherapy were termed platinum-sensitive. In contrast, patients whose disease recurred in less than 6 months were classified as platinum-resistant.

CONTACTS AND LOCATIONS:
Overall Officials: huaiwu Lu, Principal Investigator — The Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- The Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bristow RE, Tomacruz RS, Armstrong DK, Trimble EL, Montz FJ. Survival effect of maximal cytoreductive surgery for advanced ovarian carcinoma during the platinum era: a meta-analysis. J Clin Oncol. 2002 Mar 1;20(5):1248-59. doi: 10.1200/JCO.2002.20.5.1248. PMID 11870167
- [Result] Feng Z, Wen H, Jiang Z, Liu S, Ju X, Chen X, Xia L, Xu J, Bi R, Wu X. A triage strategy in advanced ovarian cancer management based on multiple predictive models for R0 resection: a prospective cohort study. J Gynecol Oncol. 2018 Sep;29(5):e65. doi: 10.3802/jgo.2018.29.e65. Epub 2018 Apr 23. PMID 30022629
- [Result] Vergote I, Coens C, Nankivell M, Kristensen GB, Parmar MKB, Ehlen T, Jayson GC, Johnson N, Swart AM, Verheijen R, McCluggage WG, Perren T, Panici PB, Kenter G, Casado A, Mendiola C, Stuart G, Reed NS, Kehoe S; EORTC; MRC CHORUS study investigators. Neoadjuvant chemotherapy versus debulking surgery in advanced tubo-ovarian cancers: pooled analysis of individual patient data from the EORTC 55971 and CHORUS trials. Lancet Oncol. 2018 Dec;19(12):1680-1687. doi: 10.1016/S1470-2045(18)30566-7. Epub 2018 Nov 6. PMID 30413383
- [Result] Suidan RS, Ramirez PT, Sarasohn DM, Teitcher JB, Iyer RB, Zhou Q, Iasonos A, Denesopolis J, Zivanovic O, Long Roche KC, Sonoda Y, Coleman RL, Abu-Rustum NR, Hricak H, Chi DS. A multicenter assessment of the ability of preoperative computed tomography scan and CA-125 to predict gross residual disease at primary debulking for advanced epithelial ovarian cancer. Gynecol Oncol. 2017 Apr;145(1):27-31. doi: 10.1016/j.ygyno.2017.02.020. Epub 2017 Feb 14. PMID 28209497
- [Result] Chereau E, Ballester M, Selle F, Cortez A, Darai E, Rouzier R. Comparison of peritoneal carcinomatosis scoring methods in predicting resectability and prognosis in advanced ovarian cancer. Am J Obstet Gynecol. 2010 Feb;202(2):178.e1-178.e10. doi: 10.1016/j.ajog.2009.10.856. PMID 20113693
- [Result] Wang J, Liu L, Pang H, Liu L, Jing X, Li Y. Preoperative PET/CT score can predict incomplete resection after debulking surgery for advanced serous ovarian cancer better than CT score, MTV, tumor markers and hematological markers. Acta Obstet Gynecol Scand. 2022 Nov;101(11):1315-1327. doi: 10.1111/aogs.14442. Epub 2022 Aug 18. PMID 35979992
- [Result] Palomar Munoz A, Cordero Garcia JM, Talavera Rubio MDP, Garcia Vicente AM, Pena Pardo FJ, Jimenez Londono GA, Soriano Castrejon A, Aranda Aguilar E. Value of [18F]FDG-PET/CT and CA125, serum levels and kinetic parameters, in early detection of ovarian cancer recurrence: Influence of histological subtypes and tumor stages. Medicine (Baltimore). 2018 Apr;97(17):e0098. doi: 10.1097/MD.0000000000010098. PMID 29702969
- [Result] Dondi F, Albano D, Bellini P, Camoni L, Treglia G, Bertagna F. Relationship between Baseline [18F]FDG PET/CT Semiquantitative Parameters and BRCA Mutational Status and Their Prognostic Role in Patients with Invasive Ductal Breast Carcinoma. Tomography. 2022 Oct 27;8(6):2662-2675. doi: 10.3390/tomography8060222. PMID 36412681